CLINICAL TRIAL: NCT06203717
Title: Cranial Electrotherapy Stimulation: Piloting a Road to PTSD Prevention in First Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: University of Rhode Island (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2091269
Record Dates: First submitted 2023-11-08; First posted 2024-01-12 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Adults
Keywords: Firefighters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Alpha-Stim AID cranial electrotherapy stimulation (Experimental): Four-week course of noninvasive cranial electrotherapy stimulation.
  Interventions: Device: Alpha-Stim AID cranial electrotherapy stimulation

INTERVENTIONS:
Device: Alpha-Stim AID cranial electrotherapy stimulation — Cranial electrotherapy stimulation using a modified square, bipolar waveform of 0.5 Hz at 100 μA to be used for four weeks on off-duty days.

SUMMARY:
The goal of this study is to test whether active duty firefighters find it possible and suitable to do cranial electrotherapy stimulation (CES) at home, and test whether CES influences measures of depression and posttraumatic stress. The main questions it aims to answer are:

* is CES feasible and acceptable in a population of firefighters, and
* does CES changes feelings of depression, anxiety, and fatigue in firefighters.

Participants will

* complete four weeks of CES at home, and
* complete daily assessments of affect and fatigue, and
* complete self-reported symptoms of depression and posttraumatic stress before and after four weeks of CES at home Participants maybe asked to
* complete an MRI scan before and after four weeks of CES at, and
* wear a device to measure their heart rate and sleep quality.

DETAILED DESCRIPTION:
Despite an urgent need for interventions that can prevent the development of posttraumatic stress disorder (PTSD) in firefighter first responders who, due to the nature of their occupation, are at ultrahigh risk for PTSD and its profound consequences, current preventative approaches suffer from low rates of efficacy or difficulties with implementation. Cranial electrotherapy stimulation (CES), a noninvasive brain stimulation technique that is FDA approved for treatment of anxiety, insomnia, and depression, offers substantial promise as a proactive preventative intervention for PTSD because of its hypothesized ability to reestablish homeostasis, a process that becomes dysregulated in individuals who develop PTSD. The proposed study is an administrative supplement that combines the unique strengths and knowledge of a complimentary team of scientists from two distinct Centers of Biomedical Research Excellence to test whether four weeks of CES is feasible and acceptable in firefighters as well as obtain early signal of CES efficacy to change subjective and objective indices of homeostatic functioning to allow a long-term collaboration with the ultimate goal to develop a safe, effective, and easily deployable intervention to prevent PTSD in first responders.

ELIGIBILITY:
Inclusion Criteria:

* Active duty firefighter in Rhode Island, USA;
* Age between 18 and 56 years old;
* Be in good medical health or, if having chronic medical conditions, these conditions needed to be stable;
* Ability to speak, read, write, and understand English sufficiently well to complete study procedures and provide informed consent.

Exclusion Criteria:

* MRI and CES-related contraindications, e.g., implanted metallic device or substances including pacemakers, cochlear implant, metallic tattoos, claustrophobia, pregnancy or planning to become pregnant during the study duration and nursing;
* Neurological conditions such as brain neoplasm, cerebrovascular events, epilepsy or history of seizures, dementia, and neurodegenerative disorders, or had previously received brain surgery;
* Report presence of suicidal ideation on QuickSCID-5 or has attempted suicide one or more times within the past twelve months;
* Exhibiting a psychiatric condition that would require inpatient or partial psychiatric hospitalization;
* Current moderate or severe alcohol or other substance abuse (excluding nicotine);
* Major or unstable medical illness requiring further investigation or treatment.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mascha van 't Wout-Frank, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.15 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Posttraumatic Stress Disorder (PTSD) Checklist for DSM-5 [Number; unit: score on PTSD Checklist for DSM-5] — Severity of posttraumatic stress symptoms as measured with the PTSD Checklist for DSM-5 (PCL-5). Scale ranges from 0 to 80 with higher scores indicating greater severity of posttraumatic stress disorder symptoms.
  score on PTSD Checklist for DSM-5 | 20
Inventory of Depressive Symptomatology-Self Report (IDS-SR). [Mean (Standard Deviation); unit: score on IDS-SR] — Presence and severity of depression symptoms assessed using the Inventory of Depressive Symptomatology-Self Report (IDS-SR). Score ranges from 0 to 84, with each of its 30 items rated on a scale from 0 to 3. Scores of 18 or above on the IDS-SR indicate the presence of clinically relevant depressive symptomatology.
  score on IDS-SR | 18.77 (11.35)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Cranial Electrotherapy Stimulation
Description: Feasibility assessed by number of completed cranial electrotherapy stimulation sessions over the course of four weeks (feasible is defined as more than 75% of sessions completed).
Time Frame: During four weeks of cranial electrotherapy stimulation at-home use
Measure: Mean (Standard Deviation); unit: percentage of CES sessions completed
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Number analyzed (Participants) | 13
percentage of CES sessions completed | 86.15 (16.51)

2. Primary Outcome: Acceptability of Cranial Electrotherapy Stimulation
Description: Acceptability assessed by number of individuals who complete at least 75% of all cranial electrotherapy stimulation sessions during four weeks
Time Frame: During four weeks of cranial electrotherapy stimulation
Measure: Count of Participants; unit: Participants
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Number analyzed (Participants) | 13
Participants | 10

3. Secondary Outcome: Severity of Symptoms of Posttraumatic Stress Disorder as Measured With the PTSD Checklist for DMS 5 (PCL-5)
Description: Score on the PTSD Checklist for DSM-5 (PCL-5). Scale ranges from 0 to 80 with higher scores indicating greater severity of posttraumatic stress disorder symptoms.
Time Frame: Post four weeks of cranial electrotherapy stimulation
Measure: Mean (Standard Deviation); unit: score on PTSD Checklist for DSM-5
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Number analyzed (Participants) | 13
score on PTSD Checklist for DSM-5 | 10.85 (10.54)
Statistical Analysis 1: Comparison: Alpha-Stim AID cranial electrotherapy stimulation; Test type: Superiority; p = 0.007, Paired-sample t-test — a priori threshold for statistical significance: p<0.05; Mean Difference (Net) = 9.15, 95% CI 2-sided [3.08 to 15.23], Standard Deviation 10.06

4. Secondary Outcome: Severity of Symptoms of Depression as Measured With the Inventory of Depressive Symptomatology-Self Report (IDS-SR)
Description: Score on the Inventory of Depressive Symptomatology-Self Report (IDS-SR). The Inventory of Depressive Symptomatology-Self Report (IDS-SR) has a total score range of 0 to 84, with each of its 30 items rated on a scale from 0 to 3. Scores of 18 or above on the IDS-SR indicate the presence of clinically relevant depressive symptomatology.
Time Frame: post four weeks of cranial electrotherapy stimulation.
Measure: Mean (Standard Deviation); unit: score on Inventory of Depressive Symptom
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
Number analyzed (Participants) | 13
score on Inventory of Depressive Symptom | 11.00 (7.54)
Statistical Analysis 1: Comparison: Alpha-Stim AID cranial electrotherapy stimulation; Test type: Superiority; p = 0.0009, Paired-sample t-test; Mean Difference (Net) = 7.77, 95% CI 2-sided [3.93 to 11.61], Standard Deviation 6.35

5. Secondary Outcome: Intensity of Feelings of Fatigue
Description: Intensity of subjective fatigue assessed once daily using a visual analog scale (VAS) with a 0 (not at all) - 100 (severe) scale.
Time Frame: Daily throughout four weeks of cranial electrotherapy stimulation
Reporting Status: Not Posted

6. Secondary Outcome: Intensity of Feelings of Anxiety
Description: Intensity of anxiety will be assessed once daily using a visual analog scale (VAS) with a 0 (not at all) - 100 (severe) scale.
Time Frame: Daily throughout four weeks of cranial electrotherapy stimulation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Weekly during the one month of at home cranial electrotherapy stimulation
Arm/Group | Alpha-Stim AID cranial electrotherapy stimulation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha-Stim AID cranial electrotherapy stimulation (N=13)
Tingling (Skin and subcutaneous tissue disorders) | 6 (6) — Tingling, itchy feeling under electrodes attached to ears
Skin redness (Skin and subcutaneous tissue disorders) | 2 (2) — Temporary skin redness under electrodes attached to ears
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 3 (3)
Mood changes (Psychiatric disorders) | 4 (4)
Difficulties concentrating (Nervous system disorders) | 0 (0)
Feeling drowsy (Nervous system disorders) | 2 (2)
Phosphenes (Nervous system disorders) | 1 (1) — Experience of brief flickering lights
Dizziness (Nervous system disorders) | 3 (3)
Nausea (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT06203717/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT06203717/ICF_001.pdf